CLINICAL TRIAL: NCT01082497
Title: Mindfulness Training and Developing the Ability of Empathy at an Inpatient Ward for Dual Diagnoses
Brief Title: Mindfulness Training for Staff (MTS)
Acronym: MTS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P REK NORD-134/2008
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Stress
Keywords: Mindfulness; Stress; Burnout; Ward atmosphere; Stress and burnout among staff, psychosocial atmosphere at the ward
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness (Experimental)
  Interventions: Behavioral: Mindfulness training
- Education (Active Comparator): 8 - weekly workshops on affect consciousness for all staff
  Interventions: Behavioral: Mindfulness training

INTERVENTIONS:
Behavioral: Mindfulness training — A course in mindfulness based stress reduction with 8 weekly group meetings and home practice between the meetings. Each meetings last for 90 minutes. Participants get workbook and cds to support home practice.
  Other Names: MBSR

SUMMARY:
The purpose of this study is to investigate whether a mindfulness based 8-week course for stress reduction, known as MBSR course, given to all staff at an inpatient psychiatric ward influences the level of stress and burnout and the psychosocial atmosphere at the ward.

The design is an intervention trial with repeated measures and control group.The focus is the interaction between unit and individuals.

All staff at both wards were invited to participate. The intervention consists of 8 weekly group meetings where the participants learn different ways of practicing mindfulness and do home practice between the meetings. The control intervention is 8 weekly workshops in affect-consciousness.

Data are collected through self-reporting questionnaires on mindfulness, work- and health-related topics at six different points. The patients at both wards answers one questionnaire about ward atmosphere at the same points.

Data wil be analyzed on SPSS statistic programme.

DETAILED DESCRIPTION:
MBSR for staff in inpatient psychiatric units

The challenges for staff working at an inpatient unit for psychotic people are many, and still more where the patients also have addiction problems. The patients are seriously ill and in need of extensive support and treatment. It is needed for the staff to be continuously aware and present, stand all kind of situations and hold out (contain) a lot of critique and threatening from the patients. Often they are too exhausted to take care of themselves and their own stress. The risk for burnout is high. The purpose of this study is to investigate whether a mindfulness based 8-week course for stress reduction, known as MBSR course, given to all staff at an inpatient psychiatric ward influences the psychosocial atmosphere at the ward.

The design of the study is an intervention trial with repeated measures and control group. The intervention consists of 8 weekly group meetings where the participants learn different ways of practicing mindfulness; sitting, walking, yoga exercises,and body scan.They are asked to practice between the group-meetings and get a workbook and cds as support.

This is a prospective intervention study with control group and repeated measures over one year follow up. The focus is the interaction between unit and individuals.

To more closely study the specific effect of mindfulness practice the control group receive an active intervention which has similarities to mindfulness practice: workshops in affect - consciousness of same amount as the MBSR-course.

All staff at the research unit and the control unit were invited to participate, each group has a number of 25 - 30 individuals. Data are collected through self-reporting questionnaires at six different points. The patients answers one questionnaire at the same points.

The inventories chosen are:

Demographics Quality of life Subjective health complains Five Facets Mindfulness Questioner (Baer) Maslach Burnout Inventory Work satisfaction Total Work load - short form Ward-atmosphere scale (also for the patients) Sick leave and number of registered harm /injury- episodes will be taken on 3 -4 points.

Hopefully this study will show that when the staff practice mindfulness this will bring about a more relaxed and accepting atmosphere followed by lesser exhaustion and anxiety. Consequences should be that mindfulness practise becomes more ordinary in psychiatric hospital wards.

ELIGIBILITY:
Inclusion Criteria:

* all staff working at the ward 50 % or more, not attending to leave during the first year.

Exclusion Criteria:

* Staff working less than 50%, planned to leave before one year.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-05; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The ability of mindfulness measured by the Five Facet Mindfulness Questionnaire | Three months before to one year follow up after the intervention
  The questionnaire measure the ability to observe, describe and act with awareness,nonreactivity and non-judgemental awareness.

SECONDARY OUTCOMES:
The amount of work stress and burnout measured with The Maslach Burnout Inventory | Three months before intervention to one year follow up after the intervention
  The questionnaire measure the dimentions emotional exchaustion,depersonalization and persomal accomplishment.

CONTACTS AND LOCATIONS:
Overall Officials: Tordis Sorensen Hoifodt, dr med. phd, Study Chair — University Hospital of North Norway
Locations (1):
- University Hospital of North-Norway, Tromsø, Troms, Norway